CLINICAL TRIAL: NCT04948450
Title: A Multidomain Intervention Program for Older People With Dementia: A Pilot Study
Brief Title: A Multidomain Intervention Program for Older People With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Geriatric Hospital (Other Government)
Responsible Party: Principal Investigator, Nguyen Xuan Thanh, Deputy Head of Palliative care department, National Geriatric Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CB1.02
Record Dates: First submitted 2021-06-04; First posted 2021-07-02 (Actual); Results first posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Dementia; Alzheimer Disease; Dementia, Mixed
Keywords: Dementia; Multidomain intervention; Older people
MeSH Terms: conditions — Dementia; Alzheimer Disease; Mixed Dementias | interventions — Social Work

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Physical activity intervention:
  Progressive resistance training (PRT) for the physical intervention will be provided at the nursing home.
  Cognitive stimulation intervention:
  The study subjects will receive cognitive intervention based on Cognitive Stimulation Therapy with rehabilitation experts.
  Social intervention:
  The social intervention will be combined with physical and cognitive interventions by doing in a group.
  Metabolic and vascular risk factors:
  Metabolic and vascular risk factors of the intervention group will be evaluated by cardiologists and endocrinologists in the study.
  Interventions: Behavioral: Physical activity intervention; Behavioral: Cognitive stimulation intervention; Behavioral: Social intervention; Other: Management of metabolic and vascular risk factors
- Control group (No Intervention): The control group will receive general health advice every 3 months based on their physical examination and blood results. They will be provided information on the vascular risk factors for dementia and will receive instruction and handouts on diet and exercise.

INTERVENTIONS:
Behavioral: Physical activity intervention — Progressive resistance training (PRT) for the physical intervention will be provided at the nursing home for 45 minutes twice a week. The sessions will be organized in groups (6-10 patients/ group) and supervised by 2 physiotherapists. Within each small group (maximum 10), participants will follow the program tailored to their individual functioning level, with constant oversight by trainers.
  People with dementia and care staff will be instructed to follow the prescribed PRT exercises for the rest of the week. Subjects will be encouraged to exercise daily.
  Arms: Intervention group
Behavioral: Cognitive stimulation intervention — The study subjects will receive cognitive intervention based on Cognitive Stimulation Therapy with rehabilitation experts. The intervention involves 14 sessions of themed activities, which typically run twice weekly. The sessions will be organized in groups (6-10 patients/ group).
  People with dementia and their care staff will be instructed on how to practice the various activities at their nursing home for the rest of the week.
  Arms: Intervention group
Behavioral: Social intervention — Social intervention will be combined with physical and cognitive interventions through doing these in a group, playing games during exercises (dancing, throwing ball to each other) or doing cognitive stimulation therapy in a group.
  Arms: Intervention group
Other: Management of metabolic and vascular risk factors — Study physicians will assess the risk of developing new chronic diseases, change in blood pressure, weight and BMI, and hip and waist circumference, blood test (glucose, lipid parameters, fasting glucose, and HbA1C if the person with dementia has diabetes) at 3 and 6 months.
  Participants in the intervention group will be provided with information on the importance of reducing risk factors, guidance on lifestyle changes and prescribing treatment if necessary by cardiologists and endocrinologists. The target for blood pressure is less than 120/90 mmHg and the target for HbA1c is less than 8 %.
  Arms: Intervention group

SUMMARY:
This is a pilot study to assess the feasibility of a multidomain intervention for older people with dementia in nursing homes. Participants will be randomized into two equal groups, to receive either an intensive multidomain intervention (intervention group) or regular health advice (control group). The intervention will include physical, cognitive, and social interventions and management of metabolic and vascular risk factors. We hypothesize that the multidomain intervention will be feasible in Vietnam, and participants who receive the intervention will show improvement in cognitive function, quality of life, behaviors, functional ability, sleep, and in reduction of falls, and death rate compared to those in the control group during the 6 months intervention period

DETAILED DESCRIPTION:
This is a two-armed, multicenter, randomized controlled pilot study, based in 3 nursing homes in Hanoi, Vietnam.

The study PI and/or researchers in the research team will contact adults aged 60 years and older in the nursing homes to introduce the study. If they are interested in participating, the study PI and/or researchers in the research team will screen them for their eligibility. If they meet the inclusion criteria and are interested in participating, written informed consent will be obtained.

Participants who agreed to participate in the study will be randomized into two equal groups, to receive either an intensive multidomain intervention (intervention group) or regular health advice (control group).

Participants in both the intervention and the control groups will be treated for dementia according to the recommendations of the Vietnam Alzheimer's Disease and Neurocognitive Disorders Association.

All participants will meet the study physician to have an examination at baseline, 3 months, and 6 months. At each examination, participants will undergo a physical examination, anthropometry (weight, hip and waist circumference), blood pressure determination, pulse rate and rhythm, risks of cardiovascular and metabolic diseases (smoking, drinking, hypertension, coronary artery disease, dyslipidemia, atherosclerosis, diabetes) and assess blood test results (lipid profile, HbA1C, and fasting glucose if patients have diabetes). Results will be provided to participants and their doctors.

In addition to what is given to both groups, participants in the intervention group will receive four intervention components: (1) physical activity intervention; (2) cognitive intervention; (3) social intervention; and (4) management of metabolic and vascular risk factors. Physical activity and cognitive stimulation interventions will be performed at separate sessions.

All outcome measures will be administered at baseline, 6 months

ELIGIBILITY:
Inclusion criteria:

We aim to enroll participants aged over 60 years old, living in nursing home, who have a diagnosis of dementia (according to DSM 5 criteria), stage mild to moderate (according to Clinical Dementia Rating scale - CDR). Participants receiving pharmacological treatment for dementia must be on a stable dose for at least 3 months prior to the study. Eligible participants must be able to mobilize independently with or without a mobility aid and without physical assistance.

Exclusion criteria are:

1. Acute and malignant diseases (e.g., advanced cancers, end-stage chronic diseases, acute myocardial infarction, stroke)
2. Symptomatic cardiovascular disease, coronary revascularization within 1 year
3. Clinical evidence of schizophrenia, severe depression, psychiatric or bipolar disorder (according to DSM-V TR criteria)
4. Alcoholism or substance dependence (according to DSM-5 criteria), currently, or within the past 2 years
5. Severe loss of vision, hearing, or communicative ability (according to the interRAI Community Health Assessment)

g. Participant or family unwilling to participate in the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anh T Nguyen, PhD, Study Director — National Geriatric Hospital; Thanh X Nguyen, MS, Principal Investigator — National Geriatric Hospital
Locations (4):
- Vietnam (4):
  - Dien Hong nursing home, Hanoi
  - National Geriatric Hospital, Hanoi
  - Nhan Ai nursing home, Hanoi
  - Orihome, Hanoi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duong S, Patel T, Chang F. Dementia: What pharmacists need to know. Can Pharm J (Ott). 2017 Feb 7;150(2):118-129. doi: 10.1177/1715163517690745. eCollection 2017 Mar-Apr. No abstract available. PMID 28405256
- [Background] Prince M, Bryce R, Albanese E, Wimo A, Ribeiro W, Ferri CP. The global prevalence of dementia: a systematic review and metaanalysis. Alzheimers Dement. 2013 Jan;9(1):63-75.e2. doi: 10.1016/j.jalz.2012.11.007. PMID 23305823
- [Background] Bich NN, Dung NTT, Vu T, Quy LT, Tuan NA, Binh NTT, Hung NT, Anh LV. Dementia and associated factors among the elderly in Vietnam: a cross-sectional study. Int J Ment Health Syst. 2019 Aug 23;13:57. doi: 10.1186/s13033-019-0314-7. eCollection 2019. PMID 31462907
- [Background] GBD 2016 Dementia Collaborators. Global, regional, and national burden of Alzheimer's disease and other dementias, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2019 Jan;18(1):88-106. doi: 10.1016/S1474-4422(18)30403-4. Epub 2018 Nov 26. PMID 30497964
- [Background] Wimo A, Guerchet M, Ali GC, Wu YT, Prina AM, Winblad B, Jonsson L, Liu Z, Prince M. The worldwide costs of dementia 2015 and comparisons with 2010. Alzheimers Dement. 2017 Jan;13(1):1-7. doi: 10.1016/j.jalz.2016.07.150. Epub 2016 Aug 29. PMID 27583652
- [Background] Fink HA, Jutkowitz E, McCarten JR, Hemmy LS, Butler M, Davila H, Ratner E, Calvert C, Barclay TR, Brasure M, Nelson VA, Kane RL. Pharmacologic Interventions to Prevent Cognitive Decline, Mild Cognitive Impairment, and Clinical Alzheimer-Type Dementia: A Systematic Review. Ann Intern Med. 2018 Jan 2;168(1):39-51. doi: 10.7326/M17-1529. Epub 2017 Dec 19. PMID 29255847
- [Background] Nguyen TA, Pham T, Dang TH, Hinton WL, Nguyen AT, Pham TL, Crotty M, Kurrle S, Bui QT, Nguyen H, Roughead EE. Towards the development of Vietnam's national dementia plan-the first step of action. Australas J Ageing. 2020 Jun;39(2):137-141. doi: 10.1111/ajag.12755. Epub 2019 Dec 9. PMID 31814244
- [Background] Streater A, Spector A, Aguirre E, Hoe J, Hoare Z, Woods R, Russell I, Orrell M. Maintenance Cognitive Stimulation Therapy (CST) in practice: study protocol for a randomized controlled trial. Trials. 2012 Jun 26;13:91. doi: 10.1186/1745-6215-13-91. PMID 22735077
- [Background] Mohs RC, Knopman D, Petersen RC, Ferris SH, Ernesto C, Grundman M, Sano M, Bieliauskas L, Geldmacher D, Clark C, Thal LJ. Development of cognitive instruments for use in clinical trials of antidementia drugs: additions to the Alzheimer's Disease Assessment Scale that broaden its scope. The Alzheimer's Disease Cooperative Study. Alzheimer Dis Assoc Disord. 1997;11 Suppl 2:S13-21. PMID 9236948
- [Background] Kivipelto M, Solomon A, Ahtiluoto S, Ngandu T, Lehtisalo J, Antikainen R, Backman L, Hanninen T, Jula A, Laatikainen T, Lindstrom J, Mangialasche F, Nissinen A, Paajanen T, Pajala S, Peltonen M, Rauramaa R, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Soininen H. The Finnish Geriatric Intervention Study to Prevent Cognitive Impairment and Disability (FINGER): study design and progress. Alzheimers Dement. 2013 Nov;9(6):657-65. doi: 10.1016/j.jalz.2012.09.012. Epub 2013 Jan 17. PMID 23332672

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: The multidomain intervention comprised: (1) physical activity; (2) cognitive intervention; (3) social intervention; and (4) management of metabolic and vascular risk factors. Physical activity and cognitive stimulation sessions were conducted separately, each held twice a week. Social intervention was integrated into the physical and cognitive intervention sessions.
  For the management of metabolic and vascular risk factors, participants received education on the importance of minimizing these risks, guidance on adopting healthier lifestyles, and treatment recommendations when necessary, provided by cardiologists and endocrinologists.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 30 | 30
Completed | 29 | 27
Not Completed | 1 | 3
Not completed — Return home | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: Multidomain intervention included: (1) physical activity; (2) cognitive intervention; and (3) social intervention as well as (4) management of metabolic and vascular risk factors. Physical activity and cognitive stimulation interventions will be performed at separate sessions
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 29 | 28 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] — Multidomain intervention included: (1) physical activity; (2) cognitive intervention; and (3) social intervention as well as (4) management of metabolic and vascular risk factors. Physical activity and cognitive stimulation interventions will be performed at separate sessions
  years
    Number | 78 (7.4) | 78 (8.8) | 78 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 9 | 10 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 30 | 30 | 60
Region of Enrollment [Number; unit: participants]
  Vietnam | 30 | 30 | 60
Severity of dementia [Count of Participants; unit: Participants]
  Mild | 11 | 11 | 22
  Moderate | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Adherence
Description: Percentageof sessions attended out of the total planned
Time Frame: 6 months
Population: Adherence was only assessed for the intervention group
Measure: Number; unit: percentage of Adherence
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 30 | 0
percentage of Adherence | 85.4 |

2. Primary Outcome: Retention
Description: The retention rate was calculated as the number (percentage) of participants in each group who did not discontinue the study.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 30 | 30
Participants | 1 | 3

3. Secondary Outcome: Global Cognition
Description: Global cognition will be measured by Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog); score ranging from 0-70, a higher score indicates worse impairment.
Time Frame: Baseline, 6 months
Population: Data were analyzed on an intention-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline | 28 (8.8) | 24.5 (8.5)
  After intervention (6 months) | 27.3 (9.5) | 29.1 (9.9)

4. Secondary Outcome: Executive Function Via Clock Drawing Test
Description: Excutive function will be assessed using Clock drawing test. Scores range from 0-10, with lower scores indicating greater cognitive impairment
Time Frame: Baseline, 6 months
Population: Data were analyzed on an intention-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline | 0.5 (1.6) | 2.3 (3)
  After intervention | 2.3 (3.4) | 2.7 (3.8)

5. Secondary Outcome: Attention Function Via Digit Span Forward
Description: Attention function will be assessed using digit span forward. Scores range from 0-12. Higher scores indicated better attention
Time Frame: Baseline, 6 months
Population: Data were analyzed on an intention-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline | 8.9 (2.5) | 9.5 (2.2)
  After intervention | 9 (2.2) | 9.1 (2.8)

6. Secondary Outcome: Atttention Function Will be Assessed Using Digit Span Backward.
Description: Higher scores indicated better attention. Scores range from 0-12. Higher scores indicated better attention
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline | 2.5 (1.5) | 2.6 (1.3)
  After intervention | 2.7 (1.5) | 3 (1.3)

7. Secondary Outcome: Behavioral and Psychological Symptoms of Dementia (BPSD)
Description: Behavioral and psychological symptoms of dementia (BPSD) will be measured using the Neuropsychiatric Inventory (NPI) questionnaire. The total NPI score ranging from 0 to 144 points. Higher scores indicate greater severity of BPSD
Time Frame: Baseline, 6 months
Population: Data were analyzed on an intention-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline | 1 (1.7) | 1 (1.9)
  After intervention | 0.8 (1.7) | 0.9 (1.7)

8. Secondary Outcome: Total Dependence of Participants Assessed Using the Barthel Index
Description: Total dependence will be assessed using the Barthel Index, with a total score of 100, where scores between 0 and 20 indicate total dependence.
Time Frame: Baseline, 6 months
Population: Data were analyzed on an intention-to-treat
Measure: Number; unit: participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 30 | 30
participants
  Total dependent (baseline) | 4 | 2
  Total dependent (After intervention) | 4 | 7

9. Secondary Outcome: Functional Ability Via the Handgrip Strength
Description: Functional ability will be assessed via the handgrip strength. Higher scores indicated better functional ability
Time Frame: Baseline, 6 months
Population: Data were analyzed on an intention-to-treat
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 30 | 30
kilograms
  Baseline | 8 (7.5) | 12.4 (14.7)
  After intervention | 12.8 (6.4) | 11.1 (6.1)

10. Secondary Outcome: Functional Ability Via 30 Seconds Sit To Stand Test
Description: Count the total number of complete stands executed in 30 seconds
Time Frame: Baseline, 6 months
Population: Data were analyzed on an intention-to-treat
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 30 | 30
events
  Baseline | 4.5 (4.2) | 3.4 (4.6)
  After intervention | 5.4 (3.9) | 1.9 (4)

11. Secondary Outcome: Fall
Description: Falls will be assessed by the fall incident report at baseline and during the study period
Time Frame: Baseline, 6 months
Population: Data were analyzed on an intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 30 | 30
Participants
  Baseline | 11 | 8
  After intervention | 6 | 7

12. Secondary Outcome: Quality of Sleep
Description: Quality of sleep will be assessed using Pittsburgh Sleep Quality Index. A global PSQI score greater than 5 distinguishing good and poor sleepers
Time Frame: Baseline, 6 months
Population: Data were analyzed on an intention-to-treat
Measure: Number; unit: participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 30 | 30
participants
  Poor sleep (baseline) | 26 | 17
  Poor sleep (after intervention) | 19 | 17

13. Secondary Outcome: Health-related Quality of Life
Description: Health-related quality of life will be assessed using the Quality of Life in Alzheimer's Disease scale. The Quality of Life in Alzheimer's Disease scale measures the overall quality of life in individuals with Alzheimer's disease. It consists of 13 items, each rated on a 4-point Likert scale. The total score is obtained by summing the scores of all 13 items, resulting in a possible range from 13 to 52 points. Higher scores indicate a better quality of life.
Time Frame: Baseline, 6 months
Population: Data were analyzed on an intention-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 30 | 30
score on a scale
  Baseline | 27.3 (4.4) | 33.6 (4.6)
  After intervention | 28.9 (4.3) | 34.4 (4.1)

14. Secondary Outcome: Death
Description: Death will be assessed through reports from care staff, nursing home records.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 30 | 30
participants | 0 | 0

15. Secondary Outcome: Functional Ability Via the Instrumental Activities of Daily Living Scale
Description: Functional ability will be assessed using the Instrumental Activities of Daily Living Scale. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women, and 0 through 5 for men.
Time Frame: Baseline, 6 months
Population: Data were analyzed on an intention-to-treat
Measure: Number; unit: participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 30 | 30
participants
  Dependent (baseline) | 26 | 29
  Dependent (After intervention) | 23 | 27

16. Secondary Outcome: Dependence of Participants Assessed Using the Instrumental Activities of Daily Living Scale
Description: Dependence will be assessed using the Instrumental Activities of Daily Living scale, which evaluates the ability to perform eight daily tasks, including using the telephone, shopping, meal preparation, housekeeping, laundry, transportation, medication management, and financial management. The total score ranges from 0 to 8, with 8 indicating full independence and scores below 8 suggesting dependence in functional activities.
Time Frame: Baseline, 6 months
Population: Data were analyzed on an intention-to-treat
Measure: Number; unit: participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 30 | 30
participants
  Dependent (baseline) | 26 | 29
  Dependent (After intervention) | 23 | 27

ADVERSE EVENTS:
Time Frame: For each participant, adverse events were collected for the duration of participation in the study (up to 6 months)
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-10-07): https://cdn.clinicaltrials.gov/large-docs/50/NCT04948450/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-07): https://cdn.clinicaltrials.gov/large-docs/50/NCT04948450/SAP_001.pdf
  • Informed Consent Form (2022-10-07): https://cdn.clinicaltrials.gov/large-docs/50/NCT04948450/ICF_002.pdf